CLINICAL TRIAL: NCT07096882
Title: Phase I Clinical Trial of SDTM001 Injection as Adjuvant Treatment for NSCLC Patients With Driver-gene-negative and Negative PD-L1 Expression After Radical Surgical Resection
Brief Title: SDTM001 Injection as Adjuvant Therapy for NSCLC Patients After Radical Surgical Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cytocraft Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDTM001-2024
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; SDT-M001; Cascade primed immune cells; CAPRI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SDT-M001 injection (Experimental)
  Interventions: Biological: SDT-M001 injection

INTERVENTIONS:
Biological: SDT-M001 injection — Cascade primed immune cells(CAPRI); SDT-M001 injection is administered at three dose levels:1.5e9 cells, 3e9 cells,6e9 cells. The cells will be reinfused in 3 divided doses, administered every other day, and the total process will take 5 days.

SUMMARY:
The goal of this clinical trial is to evaluate the safety profile and tolerability of SDT-M001 injection in NSCLC patients with driver-gene-negative and negative PD-L1 expression after radical surgical resection; to determine the recommended Phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be informed of the trial before any examinations stipulated in this trial are initiated, voluntarily sign the written informed consent form (ICF) approved by the ethics committee, and be able to comply with the research procedures.
2. Age ranges from 18 to 70 years old (including threshold), regardless of gender.
3. For participants diagnosed with primary NSCLC according to the standards of the "Chinese Medical Association guideline for clinical diagnosis and treatment of lung cancer(2024 edition)" and the "Clinical Practice Guideline for Primary Lung Cancer(2022 Version)", and who have undergone radical surgical resection (R0) treatment, the TNM stage is classified as stage IIA - IIIB according to the American Joint Committee on Cancer staging system(AJCC),9th edition.
4. There is no disease recurrence (including local recurrence) after radical surgical resection (R0) treatment, and the estimated time of apheresis is within one year after the operation.
5. Previous tests for driver gene mutations (e.g., EGFR, ALK) were negative, and PD-L1 expression in tumor tissues was negative as detected.
6. Platinum-based chemotherapy (one to four cycles) has been completed before screening.
7. The ECOG performance status score is ≤1 point, the expected survival time is ≥12 months, and follow-up can be conducted as stipulated in the protocol.
8. Major organ functions must be normal (no corrective treatment with any blood components, cell growth factors, or albumin infusion within 14 days before obtaining laboratory tests) and meet the following requirements: White blood cells (WBC) ≥3.5×109 cells/L, lymphocytes (LYM) ≥0.8×109 cells/L, platelets (PLT) ≥80×109 cells/L, absolute neutrophil count ≥1.5×109 cells/L, hemoglobin ≥90g/L; Total bilirubin ≤1.5×upper limit of normal value (ULN), alanine aminotransferase (ALT) ≤2.5×ULN, aspartate aminotransferase (AST) ≤2.5×ULN; Creatinine ≤1.0×ULN, or creatinine clearance rate ≥60mL/min (using the Cockcroft-Gault method); International Normalized Ratio (INR) ≤1.5.
9. Participants must have sufficient venous access for the apheresis.
10. Eligible participants with fertility (both male and female) must agree to use reliable contraceptive methods (hormones or barrier methods or abstinence) during the trial and for at least one year after the last reinfusion of SDTM001 injection; Female participants within childbearing age must have a negative pregnancy blood test within 7 days prior to enrollment; Male participants were not allowed to donate sperm from the first infusion to one year after the last infusion.

Exclusion Criteria:

1. Participants who have participated in other clinical trials of investigational agents or devices for therapeutic intent within 4 weeks prior to screening.
2. Participants who have received cancer treatment such as chemotherapy, radiotherapy, biological therapy, targeted therapy, or immunotherapy within 4 weeks prior to screening.
3. Participants who underwent gene-modified anti-tumor immune cell therapy (e.g., CAR-T cells, CAR-NK cells) within one year or non-gene-modified therapy (e.g., NK cells, DC cells, DC-CIK cells) within half a year prior to screening.
4. Participants with impaired cardiac function or significant cardiovascular diseases, including any of the following:

(1) Acute myocardial infarction or unstable angina pectoris ≤6 months prior to screening; (2) New York Heart Association classified III/IV congestive cardiac failure; (3) Uncorrected severe arrhythmia and hypertension ≥150/100 mmHg; (4) Prolonged QTc interval (> 450ms in males , > 470ms in females); (5) History of other significant cardiovascular diseases (e.g., valve replacement surgery, coronary artery bypass grafting).

5. Participants with a history of drug addiction, alcoholism (defined as average daily pure alcohol intake ≥61g for men or ≥41g for women), or substance abuse.

6. Participants with systemic active infections requiring treatment, including but not limited to HIV-positive, syphilis positive, or clinically active hepatitis A/B/C infection.

7. Participants with severe autoimmune diseases or immunodeficiency, such as those requiring long-term (≥2 months) systemic immunosuppressant (e.g., steroid) for severe autoimmune diseases, or those with severe immune-mediated symptomatic diseases (e.g., ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune vasculitis(e.g., Wegener granulomatosis)).

8. Participants who require systemic immunosuppressants (e.g., cortisol, hydroxyurea) within 28 days prior to screening or during the trial, or other immunomodulators (e.g., interferon-alpha/gamma, GM-CSF, mTOR inhibitors, cyclosporine, thymosin).

9. Participants with a history of organ transplantation, allogeneic stem cell transplantation or renal replacement therapy; 10. Participants who have received live vaccines within 28 days prior to screening or plan to receive live vaccines during the study period.

11. Participants who have undergone major operations within 4 weeks prior to screening.

12. Participants with known allergic reactions to SDT-M001 injection, its active ingredients, excipients, or a history of allergy to cell products 13. Participants with a history of or current other malignant tumors, except:

1. Malignant tumors with no recurrence for ≥5 years after radical treatment
2. Cured cervical cancer or breast carcinoma in situ, basal cell carcinoma or squamous cell carcinoma.

14. Participants with any mental illness or severe mental disorder (e.g., dementia, altered mental status) that may affect informed consent or comprehension of questionnaires.

15. Breastfeeding women are excluded. 16. Participants who are deemed by the investigator to be unable to complete trial visits, evaluations, or follow-ups, have poor compliance, or are otherwise unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-07-26 (Estimated); Primary Completion 2027-06-26 (Estimated); Study Completion 2029-06-26 (Estimated)

PRIMARY OUTCOMES:
Safety profile of SDT-M001 injection | From enrollment up to 24 Months After the end of the last infusion
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards. Adverse events (AE) of all subjects entering this trial, including serious adverse events (SAE); laboratory examination indicators.
Tolerability of SDT-M001 injection | From enrollment to 28 days after the end of the last infusion
  The number and severity of dose-limiting toxicity (DLT) events. Calculate the incidence of DLT.
RP2D | Until the end of the study
  If the maximum tolerated dose (MTD) has been proven to be feasible for long-term clinical administration in a reasonable number of subjects, then this dose is usually RP2D.

SECONDARY OUTCOMES:
Therapeutic effect evaluation | From enrollment up to 24 Months After the end of the last infusion.
  Efficacy evaluation will be conducted according to the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China